CLINICAL TRIAL: NCT00632580
Title: Intraartikulær Versus ekstraartikulær Bolus Injektion Med Ropivacain Ved Total knæalloplastik: et Prospektivt, Randomiseret, Dobbeltblindet, Kontrolleret Studie
Brief Title: Intra- Versus Extraarticular Injection of Ropivacaine in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Hvidovre University Hospital, Department of Anesthesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-D-2007-0079
Record Dates: First submitted 2008-02-28; First posted 2008-03-10 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Injections, Intra-Articular; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): intraarticular injection with local anesthetic
  Interventions: Drug: intraarticular injection with ropivacaine
- 2 (Experimental): intracapsular injection with local anesthetic
  Interventions: Drug: extraarticular injection with ropivacaine

INTERVENTIONS:
Drug: intraarticular injection with ropivacaine
  Arms: 1
Drug: extraarticular injection with ropivacaine
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the optimal site for application of local anesthetics in total knee arthroplasty surgery. The hypothesis is, that improved pain relief is obtained when administering local anesthetics in the tissues sourrounding the knee joint compared to the knee joint itself.

ELIGIBILITY:
Inclusion Criteria:

* eligible for elective total knee arthroplasty
* able to speak and understand Danish
* able to give informed consent

Exclusion Criteria:

* alocohol or medical abuse
* allergies to local anesthetics
* age < 18 yrs.
* intolerance to opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
pain | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Andersen, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Denmark